CLINICAL TRIAL: NCT06905808
Title: E-Sense® Normal Values of Urodynamic Pressures Using E-Sense® Catheters
Acronym: ESNS-01
Status: Not yet recruiting | Type: Observational
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-00085
Record Dates: First submitted 2025-03-18; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Lower Urinary Track Symptoms; Urodynamic Exam
Keywords: Urodynamic; Lower Urinary Track Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects indicated for UDS study: The e-Sense® catheters will be used in all subjects to assess primary and secondary objectives. It is a single arm study with no comparative, placebo, sham or control arm.
  Interventions: Device: eSense 7Fr Single Sensor Bladder Catheter

INTERVENTIONS:
Device: eSense 7Fr Single Sensor Bladder Catheter — Urinary and abdominal catheters inserted into the body to measure pressure for urodynamics.
  Other Names: eSense 7Fr Abdominal Catheters, eSense 7Fr Dual Sensor Urethral Catheters

SUMMARY:
In this post-market observational study, subjects referred to urodynamic testing will be approached to enroll in a clinical study to define the normal range of pressure values utilizing e-Sense® catheters. Urodynamic test results using the study devices will be provided back to the study sponsor for test interpretation and to publish. The urodynamic information collected using the study devices will be used in the UDS test interpretation for each subject enrolled, unless there is a reason to believe the test should be repeated (i.e. inconclusive results).

DETAILED DESCRIPTION:
Subjects who are referred to undergo a Urodynamics will be recruited to participate. Initial resting pressures will be measured/recorded using the e-Sense® and water-filled catheter (dual-catheterized) in lying, sitting, and standing positions for each subject. The study will collect various urodynamic pressure values at regular intervals during bladder filling. The detrusor pressures before filling will then be compared with the pressures collected during bladder filling to determine normal pressure value ranges. Urethral pressures will also be measured using e-Sense® and water-filled catheters, and the values compared. The goal is to provide users of the e-Sense® catheter as to what values should be expected when good quality measurements are being made.

ELIGIBILITY:
Inclusion Criteria:

* Subjects medically indicated for Urodynamic procedure between ages 20-35 or > 50 years old (equally split male and female)
* Due to aging and giving birth significantly affecting the urethra:
* Female subjects 20-35 should be nulliparous.
* Female subjects > 50 years old should have given birth to at least one child vaginally. Further caesarian births would not mean exclusion from the study.
* Subjects with range of BMI values
* Subject provides written authorization and/or consent per institution or geographical requirements

Exclusion Criteria:

* Subjects with cognitive or psychiatric conditions that interfere with or precludes direct and accurate communication regarding the study, giving informed consent
* Any anal / rectal symptoms and/or surgery
* Pregnant women
* Subjects with active untreated bladder infections (not including patients with asymptomatic bacteruria)
* Subjects having greater than 300 mL post void residual on the clinic visit uroflowmetry test

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are medically indicated to receive a Urodynamic Procedure in the UK
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the range of normal pressure values for different patient positions measured by the e-Sense® catheter | Periprocedural, during Urodynamic Procedure
  The primary endpoint will be measured by recording the subject in three different positions (sitting, lying and standing) to determine a range normal pressures value. The values will be recorded on each subject case report form.

SECONDARY OUTCOMES:
To compare pressure values measured by the e-Sense® catheters to the pressures simultaneously measured via a separate water filled catheters. | Periprocedural, during Urodynamic Procedure
  To investigate the change of pressures readings when the subject changes positions, a comparison would be made in the change of pressure recorded by both e-Sense® and water filled catheters when the subject moves from supine to sitting and from sitting to standing.

IPD SHARING:
Plan to Share IPD: Undecided